CLINICAL TRIAL: NCT01276769
Title: Phase IIb Trial of Paclitaxel Plus Carboplatin Versus Paclitaxel Plus Epirubicin as Neoadjuvant Treatment in Locally Advanced Triple-negative Breast Cancer
Brief Title: Comparison Study of Neoadjuvant Paclitaxel Plus Carboplatin/Epirubicin Treatment in Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, ZHANG Pin, Medicine Oncology Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2010A03
Record Dates: First submitted 2010-12-10; First posted 2011-01-13 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Neoadjuvant chemotherapy; Platinum
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ET (Active Comparator): The control arm receive the paclitaxel plus epirubicin
  Interventions: Drug: Paclitaxel and epirubicin
- PC (Experimental): the experimental arm which receive the paclitaxel combined with carboplatin
  Interventions: Drug: Paclitaxel plus carboplatin

INTERVENTIONS:
Drug: Paclitaxel plus carboplatin — Paclitaxel 175 mg/m2 D1 i.v., carboplatin AUC=5 D2 i.v.
  1 cycle = 21days 2-6cycles
  Arms: PC
Drug: Paclitaxel and epirubicin — Paclitaxel 175 mg/m2 D3 i.v.,Epirubicin 75mg/m2 D1，2 i.v.
  1 cycle = 21days
  2-6cycles
  Arms: ET

SUMMARY:
This study is to compare the effective of Paclitaxel combined with Epirubicin and Paclitaxel plus Carboplatin in the neoadjuvant treatment for TNBC. And the investigators hypothesized that paclitaxel combined with carboplatin is more sensitive to TNBC compared with Paclitaxel plus Epirubicin,this study will also have a look into the relation of BRCA1 mutation and sensitive to carboplatin.

DETAILED DESCRIPTION:
It is know that triple-negative breast cancer(TNBC) is more aggressive than non-triple negative breast cancer in both pathological features and clinical prognosis,and there is no standard chemotherapy regimens especially for TNBC. NCCN guidelines recommends Paclitaxel or Epirubicin based regimens as the preferred regimens both for the adjuvant chemotherapy and the treatment of Recurrence and Metastatic breast cancer.The combination of these two drugs is considered as a strong arrangement and therefore,is common used in Triple negative breast cancer patients because of its poor prognosis.

According to the results of some retrospective studies, platinum-based chemotherapy regimens showed a promising sensitive to Triple negative breast cancer patients compared with regimens without platinum.

This study is to compare the effective of Paclitaxel combined with Epirubicin and Paclitaxel plus Carboplatin in the neoadjuvant treatment for TNBC. And the investigators hypothesized that paclitaxel combined with carboplatin is more sensitive to TNBC compared with Paclitaxel plus Epirubicin,this study will also have a look into the relation of BRCA1 mutation and sensitive to carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 18 to 70 years;
* WHO Performance status (ECOG) of 0 or 1
* Core biopsy histologically proven Ⅱa-Ⅲc phase breast cancer (regardless of the type);
* Immunohistochemisty（IHC）：ER-，PR-，CerB2-；Triple negative （ER-PR-Her-2-） Hormone receptor negativity is defined as ER<10%, PR<10% (IHC), HER2 negativity is defined as IHC 0-1+, or [IHC 2+ and FISH or CISH negative]；
* Adequate hematological function (neutrophil count ³ 2x109/l, platelet count ³ 100x 109/l, Hemoglobin > 9 g/dl);
* Adequate hepatic function: ASAT and ALAT £ 1.5 ULN alkaline phosphatases £ 2.5 ULN,total bilirubin £ 1,5 ULN;
* Adequate renal function: serum creatinine £ 1.5 ULN;
* Adequate cardiac function, LEVF value > 50% by Muga scan or echocardiography，and electrocardiogram doe not show specific abnormality；
* Patients accepting contraception intake during the overall length of treatment if of childbearing potential;
* Signed written informed consent.

Exclusion Criteria:

* Any tumor ³ T4a (UICC1987) (cutaneous invasion, deep adherence, inflammatory breast cancer);
* ER+ or PR+ or Her-2 overexpression
* Any chemotherapy, hormonal therapy or radiotherapy before
* Previous cancer in the preceding 10 years;
* Patients already included in another therapeutic trial involving an experimental drug;
* Patients with other concurrent severe and/or uncontrolled medical disease or infection which could compromise participation in the study;
* LEVF < 50% (MUGA scan or echocardiography);
* Clinically significant cardiovascular disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension (>150/90), myocardial infarction or cerebral vascular accidents) within 6 months prior to chemotherapy;
* Known prior severe hypersensitivity reactions to agents that will be received;
* Women who are pregnant or breastfeeding. Adequate birth control measures should be taken during study treatment phase;
* Women with a positive pregnancy test en enrollment or prior to study drug administration;
* Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Individual deprived of liberty or placed under the authority of a tutor.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Pathology of specimens derived from the breast modified radical mastectomy/Breast-conserving surgery | One week after the surgery
  After patients complete the neoadjuvant chemothreapy and receive the surguries,we can get their pathology ，and compare the pCR（pathological complete remission）rates of two amrs

SECONDARY OUTCOMES:
follow-up the patient every 3-6 months to obtain the 3 year-DFS(disease free survival ) and OS(overall survival ) | we follow up the patients every 6 month ,up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: ZHANG Pin, BD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer institute &Hospital，Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China